CLINICAL TRIAL: NCT05214729
Title: Diagnostic Performance of a Net Ultrafiltration Challenge to Predict Preload Dependence in Critically Ill Patients Under Continuous Renal Replacement Therapy
Brief Title: A Net Ultrafiltration Challenge to Predict Preload-dependence (UF CHALLENGE)
Acronym: UF CHALLENGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL21_1250; 2021-A02939-32 (Other: ID RCB)
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; renal replacement therapy; hemodynamics; preload dependence; net ultrafiltration
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast to Slow Group (Experimental): The Fast to Slow Group corresponds to enrolled patients randomized, following the sequential crossover design, to first perform the fast UF challenge immediately after inclusion, followed by the slow UF challenge after a washout period of 24 hours.
  Interventions: Diagnostic Test: Fast ultrafiltration challenge; Diagnostic Test: Slow ultrafiltration challenge
- Slow to Fast Group (Experimental): The Slow to Fast Group corresponds to enrolled patients randomized, following the sequential crossover design, to first perform the slow UF challenge immediately after inclusion, followed by the fast UF challenge after a washout period of 24 hours.
  Interventions: Diagnostic Test: Fast ultrafiltration challenge; Diagnostic Test: Slow ultrafiltration challenge

INTERVENTIONS:
Diagnostic Test: Fast ultrafiltration challenge — The fast ultrafiltration challenge will be performed once in all enrolled participants, in the order defined by randomization. The fast ultrafiltration challenge consists of the net removal of 250 ml of ultrafiltrate by setting net ultrafiltration rate to 1000 ml/h, applied for 15 minutes. The cardiac output will be measured before and after the UF challenge, by mean of the transpulmonary thermodilution technique, and its relative variation from baseline will be quantified to evaluate the impact of the UF challenge on cardiac preload.
  The UF challenge will be preceded and immediately followed by a postural change maneuver to assess the presence or absence of preload dependence. The postural change maneuver is positive in case of a +10% variation in continuous cardiac index over 1 minute, and is considered as the reference diagnostic test to which UF challenge diagnostic performance will be compared.
Diagnostic Test: Slow ultrafiltration challenge — The slow ultrafiltration challenge will be performed once in all enrolled participants, in the order defined by randomization. The slow ultrafiltration challenge consists of the net removal of 250 ml of ultrafiltrate by setting net ultrafiltration rate to 500 ml/h, applied for 30 minutes. The cardiac output will be measured before and after the UF challenge, by mean of the transpulmonary thermodilution technique, and its relative variation from baseline will be quantified to evaluate the impact of the UF challenge on cardiac preload.
  The UF challenge will be preceded and immediately followed by a postural change maneuver to assess the presence or absence of preload dependence. The postural change maneuver is positive in case of a +10% variation in continuous cardiac index over 1 minute, and is considered as the reference diagnostic test to which UF challenge diagnostic performance will be compared.

SUMMARY:
Hemodynamic instability episodes are a frequent complication of renal replacement therapies in critically ill patients, and their incidence is associated with worse survival. Hypovolemia, identified by the existence of biventricular preload dependence, is responsible for one episode out of two, and may justify a decrease in or cessation of fluid removal by net ultrafiltration (UF). To date, preload dependence is most frequently identified by evaluating the effects on cardiac output of postural changes (passive leg raising), impact of cardio-pulmonary interactions in ventilated patients, or fluid challenge. However, none of these tests may help identify a patient whose cardiac output is at risk of becoming preload dependent, that is situated at the inflexion point of the Frank Starling curve.

Our study aims to evaluate the effects on cardiac output (measured by a transpulmonary thermodilution technique) of 2 net ultrafiltration challenges, consisting fast removal of 250 ml of ultrafiltrate over 15 and 30 minutes respectively, and compare their diagnostic performance to the reference technique of preload dependence assessed by postural changes (passive leg raising) performed after the UF challenge.

Enrolled participants will undergo both UF challenges, following a randomized crossover design, in which the order of UF challenge duration (15 or 30 minutes) is randomized, separated by a washout period of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* adult patient, aged 18 year or older
* under mechanical ventilation and continuous general anesthesia, with a positive end-expiratory pressure of 5 cmH2O or more
* with stage 3 KDIGO acute kidney injury
* treated with continuous renal replacement therapy for less than 14 days
* ongoing continuous cardiac output monitoring
* with a predicted intensive care length of stay of 24 hours or more at time of screening

Exclusion Criteria:

* High arterial lactate concentration, > 4.0 mmol/L at time of screening
* Calibrated cardiac index < 2.0 L/min/m2 or > 4.0 L/min/m2 at time of screening
* Positive postural change maneuver in the last 2 hours preceding screening
* Patient under extracorporeal membrane oxygenation
* Patient with active bleeding requiring emergent transfusion
* Patient under chronic maintenance dialysis or renal transplant recipient
* Acute ischemic or hemorrhagic stroke complicated with coma and requiring mechanical ventilation
* Fulminant hepatitis (acute liver injury, hepatic encephalopathy, icterus and a drop in prothrombin < 50% in less that 15 days
* Impossible postural change maneuver
* Pregnant or lactating patient
* Imminent death
* Patient under legal protection measures as by French regulation
* Patient already enrolled in the present study
* Patient already participates in a study with protocolized net ultrafiltration, ongoing at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
UF challenge diagnostic performance to identify preload dependence risk, evaluated by the area under the curve of the receiver-operating characteristic curve (ROC) of the relative cardiac output variation | The relative variation in cardiac output induced by UF challenges is quantified immediately at the end of UF challenges. The postural maneuver is performed immediately after the end of UF challenges.
  The discriminatory performance of the relative variation in cardiac output (in %) between baseline and after the UF challenge will be quantified using the ROC, using the result of the postural change maneuver (negative or positive) performed after the UF challenge as the reference binary classifier. A 95% confidence interval of the ROC will be computed, as well as its statistical significance, as compared to a random guess, using the Delong method.

SECONDARY OUTCOMES:
Respective diagnostic performances of slow and fast UF challenges to identify preload dependence risk, evaluated by their respective ROC of the relative cardiac output variation. | The relative variation in cardiac output induced by UF challenges is quantified immediately at the end of UF challenges. The postural maneuver is performed immediately after the end of UF challenges.
  The discriminatory performance of the relative variation in cardiac output (in %) between baseline and after each UF challenge (slow and fast) will be quantified using the ROC, using the result of the postural change maneuver (negative or positive) performed after the UF challenge as the reference binary classifier. A 95% confidence interval of the ROC will be computed, as well as its statistical significance, as compared to a random guess, using the Delong method.
Optimal threshold value of the relative cardiac output variation (in %) following a UF challenge | The relative variation in cardiac output induced by UF challenges is quantified immediately at the end of UF challenges.
  using the ROC of the relative cardiac output variation induced by UF challenges, an optimal cutoff value will be determined, using the Youden method. This optimal threshold will allow the associated parameters describing its diagnostic performance: sensitivity, specificity, positive and negative predictive values, likelihood ratios.
UF challenge diagnostic performance to identify pre-existing preload dependence, evaluated by the ROC of the relative cardiac output variation. | The relative variation in cardiac output induced by UF challenges is quantified immediately at the end of UF challenges. The postural maneuver is performed immediately before UF challenges.
  The discriminatory performance of the relative variation in cardiac output (in %) between baseline and after the UF challenge will be quantified using the ROC, using the result of the postural change maneuver (negative or positive) performed before the UF challenge as the reference binary classifier. A 95% confidence interval of the ROC will be computed, as well as its statistical significance, as compared to a random guess, using the Delong method.
Comparison of slow and fast UF challenge diagnostic performance, using their respective ROC of relative cardiac output variation. | The relative variation in cardiac output induced by UF challenges is quantified immediately at the end of UF challenges.
  Statistical comparison of slow and fast UF challenges ROCs will be performed using the Delong methods
Impact of UF challenges on hemodynamics: central venous pressure (mmHg), heart rate (bpm), mean and pulse arterial pressures (mmHg), extravascular lung water (ml/kg), vascular permeability, and global end diastolic volume (ml/kg). | The variation in hemodynamic parameters induced by UF challenges is quantified immediately at the end of UF challenges.
  Each parameter will be evaluated individually, and its absolute and relative variations from baseline reported. The respective effect of slow and fast UF challenges will also be compared, using mixed effects models, accounting for the repetition of measurements in enrolled patients.
Association of UF challenges with hemodynamic instability, quantified by the elapsed time between the UF challenge and the occurrence of first hemodynamic instability episode, censored at 8 hours. | Censor time at 8 hours after the end of the UF challenge. This evaluation and time frame is applied twice, after each UF challenge in all enrolled patients.
  Following UF challenges, and over the 8 following hours, we will record all following hemodynamic events: mottles appearance or extension, de novo tachycardia > 120 bpm, de novo arterial hypotension (defined as a mean arterial pressure < 65 mmHg requiring immediate clinical intervention), or de novo cardiac output drop (defined as a decrease > 15% or below 2.2 L/min/m2). The time to event will be analyzed using a Cox mixed effects regression model, adjusted for patient severity of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BITKER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Department of Intensive Care, Croix Rousse hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biscarrat C, Deniel G, Chivot M, Yonis H, Chauvelot L, Mezidi M, Richard JC, Bitker L. Diagnostic performance of a 250-ml net ultrafiltration challenge to identify risk of preload-dependence in critically ill patients undergoing continuous renal replacement therapy: a randomized, cross-over trial. Crit Care. 2025 Oct 21;29(1):446. doi: 10.1186/s13054-025-05674-3. PMID 41121412